CLINICAL TRIAL: NCT03916913
Title: Tyrosine Kinase Inhibitor Followed by Thoracic Radiotherapy for Stage IV EGFR Mutant Non-small Cell Lung Cancer: A Phase II Clinical Trial
Brief Title: TKI Followed by Thoracic Radiotherapy for Stage IV EGFR Mutant NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jingbo Wang, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201805002
Record Dates: First submitted 2019-04-13; First posted 2019-04-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
Keywords: Non small cell lung cancer; Oligo-metastasis; EGFR activating mutation; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local therapy (Experimental): Consolidation local radiotherapy
  Interventions: Radiation: Local radiation therapy

INTERVENTIONS:
Radiation: Local radiation therapy — Local radiotherapy on all sites of disease including primary and metastatic lesions

SUMMARY:
In this phase II trial with single arm, we aim to investigate the clinical efficacy and toxicity profile of local radiotherapy on all disease sites for EGFR-mutant oligo-metastatic NSCLC (no more than 3 metastatic lesions) who did not experience disease progression after at least 3 months of TKI therapy.

DETAILED DESCRIPTION:
Tyrosine kinase inhibitor (TKI) has been widely accepted as the first-line therapy for stage IV NSCLC with active mutation of EGFR. Olio-metastasis is a disease status between localized and extended status of disease, namely with the limited number of lesions, which is generally defined as ≤ 5. A couple of phase II studies have shown that consolidation local management was able to prolong the local-regional tumor control and might further improve overall survival (OS) for oligo-metastatic NSCLC who have gained disease control from systemic therapy. However, there is lack of data regarding whether local radiotherapy (RT) could improve progression free survival (PFS) and OS for NSCLC with active EGFR mutation who have benefited from TKI. In this phase II trial with single arm, we aim to investigate the clinical efficacy and toxicity profile of local radiotherapy on all disease sites for EGFR-mutant oligo-metastatic NSCLC (no more than 3 metastatic lesions) who did not experience disease progression after at least 3 months of TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75;
* ECOG performance status 0-1;
* Patients must provide study specific informed consent prior to study entry;
* Pathologically or cytologically diagnosed as NSCLC;
* EGFR activating mutation to TKI approved by histology, cytology or circulation tumor DNA;
* Stage IV NSCLC with ≤ 3 metastatic lesions (AJCC, 8th ed.) confirmed by meticulous radiographic examination. Brain MRI and 18F PET/CT is strongly recommended unless there is a contraindication;
* Patients have received≥3 months of TKI therapy and do not received disease progression;
* HB ≥ 10.0 g/dL;
* Absolute number of neutrophil granulocyte ≥ 1.5 × 109/L;
* Absolute number of PLT ≥ 100 × 109/L;
* Total bilirubin ≤ 1.5 folds of the maximum extent;
* ALT and AST ≤ 2.0 folds of the maximum extent;
* Cr ≤ 1.25 folds of the maximum extent and Ccr ≥ 60mLl/min.

Exclusion Criteria:

* Patients have received thoracic radiotherapy before;
* Malignant pleural effusion, pericardial effusion or peritoneal effusion;
* Patients have severe pulmonary comorbidity, such as ILD, COPD or other active pulmonary disease;
* Any unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, CHF (NYHA ≥ II), MI within 6 months of enrollment, severe arrhythmia requiring medication，hepatic, nephric or metabolic disease;
* HIV infection；
* Pregnancy or lactation women;
* ECOG status ≥2；
* Mixed SCLC component;
* Other factors that is considered ineligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  Duration between the first date of TKI administration and disease progression or last follow-up

SECONDARY OUTCOMES:
Overall response | 1 month after RT
  Post-RT response compared with the baseline status at the first data of TKI administration
Overall survival | 2 year
  Duration between the first date of TKI administration and any cause of death or last follow up
Time to progression of initial lesions | 1 year
  Duration between the first date of TKI administration and the progression of the initial lesions or last follow up
Time to appearance of new metastatic lesions | 1 year
  Duration between the first date of TKI administration and the occurrence of new lesions or last follow up
Treatment related toxicity | 1 year
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
EORTC Quality of life | 1 year
  Quality of life evaluation using EORTC questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, MD, Principal Investigator — Cancer Hospital, CAMS
Locations (1):
- Cancer Hospital/Institute, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No